CLINICAL TRIAL: NCT01774916
Title: Identification of Genetic and Cellular Markers Associated With Vascular Endothelial Modifications in Cutaneous Arteriovenous Malformations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2012-A00893-40; 2012-26 (Other: AP HM)
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Cutaneous Arteriovenous Malformations
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients (Other)
  Interventions: Genetic: blood samples
- volunter (Other)
  Interventions: Genetic: blood samples

INTERVENTIONS:
Genetic: blood samples

SUMMARY:
Cutaneous Arteriovenous malformations (AVM's) rare congenital high-flow vascular malformations in which arteries and veins are directly connected through a complex web of abnormal arteries and veins instead of a normal capillary network. Arterial feeders and enlarged draining veins directly connect through arteriovenous fistulas that create the "nidus". The natural history of AVMs is organized into a clinical staging system: during the first phase of quiescence, the arteriovenous malformation mimics a capillary malformation. After many years, the AVM may enlarge with loco-regional expansion and tissular destruction. At the ultimate stage, AVM may impact the heart function. They are considered non malignant but can expand and become a significant clinical risk when extensive. The management of these high flow AVM remains often problematic. Complete and large surgical excision of the nidus after hyperselective embolization is the only potential therapeutic solution but this, is often difficult if not impossible. There is no pathogenetic hypothesis for the development of these malformations. Histopathological examination (performed only on surgical resection specimen) is poor and does not provide sufficient evidence to assess the evolutivity or the severity of the MAV. Recent data hypothesize that these vascular malformations are associated with alterations of the vascular endothelium caused by genetic abnormalities involved in the control of angiogenesis and vascular homeostasis. The detection of these anomalies allows the search for cellular and genetic markers that might be useful to optimize the clinical classification, staging, predicting the evolution of these defects and some understanding of its pathophysiological mechanisms. To our knowledge, no studies to identify cellular markers / genetic and endothelial associated with the development of cutaneous AVMs have been published to date.

ELIGIBILITY:
Inclusion Criteria:

* Male or feminine Subject
* Subject of 10 and more years old,
* Subject weighing more than 55 kg. patients:
* Subject presenting a cutaneous artério-venous deformation there outside of any other deformation or known vascular tumor.
* Subject presenting no other susceptible pathology to influence endothéliaux markers (Renal insufficiency, inflammatory pathology chronicles, infections, pathologies cardiovascular, diabetes, evolutionary tumoral pathology).

volunteers:

* Unhurt Subject of deformation or vascular tumor.
* Subject presenting no other susceptible pathology to influence endothéliaux markers(scorers) (Renal insufficiency, inflammatory pathology chronicles, infections, pathologies cardiovascular).

Exclusion Criteria:

* Subject of less than 10 years old
* Subject weighing less than 55 kg
* Subject presenting another type(chap) of vascular vascular deformation or tumor

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The exploration of the microparticles, endothelial cells and progenitor cells | 36 months

SECONDARY OUTCOMES:
investigate the relationship between endothelial markers and genetic and clinical characteristics of the disease | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: michele DAMON, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France